CLINICAL TRIAL: NCT06907706
Title: Active Living After Cancer: Implementation Within Be Well Acres Homes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0231
Record Dates: First submitted 2025-03-14; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Fatigue
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Exercise; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives the ALAC intervention following the baseline assessment
  Interventions: Behavioral: Physical Activity/Physical Functioning; Behavioral: Quality of Life
- Waitlist Control (Active Comparator): Receives the ALAC intervention following the 3-month assessment
  Interventions: Behavioral: Physical Activity/Physical Functioning; Behavioral: Quality of Life

INTERVENTIONS:
Behavioral: Physical Activity/Physical Functioning — The physical activity portion of the program sessions focuses on teaching cognitive and behavioral skills to increase physical activity, including goalsetting, self-monitoring, overcoming barriers to physical activity, enlisting social support, and how to handle "high risk" situations that may result in relapses to a sedentary lifestyle. The health educator teaches participants about various forms of moderate intensity activity and has them practice brief bouts of activity of various types to ensure that they are doing the activities safely and correctly. Each week participants receive a handout to provide information about the behavioral skill taught that week. The program also provides activity trackers (week 1) and resistance bands (week 5). The pedometer assists participants in self-monitoring their activity, and the resistance bands provide a form of home-based exercise that participants can do even with limited space.
Behavioral: Quality of Life — The survivorship portion of the program features a guided discussion on a different topic each session. The goals of the discussion are to present information about the topic, answer participants' questions about the topic, encourage participants to share solutions and ideas relevant to the topic with each other, and provide information on community resources participants can access if they require additional help. The health educator makes a brief presentation about the topic, answers questions, and then asks a series of 2-3 open-ended questions to facilitate discussion about the topic. At the end of the session, the health educator navigates participants who need additional information or service related to the topic to resources in the community.

SUMMARY:
The goal of this research study is to learn more about a physical activity program adapted for cancer survivors.

DETAILED DESCRIPTION:
Primary Objectives:

Evaluate the effectiveness of ALAC adapted for delivery in Acres Homes, using a randomized wait- list-control group design. The primary outcome will be physical functioning as measured by the 30- second sit-to-stand test at 12 weeks. Secondary outcomes will include physical functioning measured by the six-minute walk, objective and self-reported physical activity, social connectedness, and quality of life. The investigators will also investigate whether program effects are maintained at 6 months. Hypothesis: Cancer survivors in the adapted ALAC program will increase their physical activity and improve their physical functioning from baseline to the end-of-intervention assessment, compared to a wait-list-control group.

Compare the reach of the ALAC program in Acres Homes to ALAC in other persistent poverty neighborhoods in Houston. Hypothesis: The Acres Homes adaptation of ALAC will have a greater reach (percent of cancer survivors enrolling in ALAC in a specific neighborhood) than in other persistent poverty neighborhoods in Houston.

Explore the moderating effects of social and environmental variables on program effectiveness. Hypothesis 3A:Participants' financial distress, experiences of discrimination, health literacy, and social connectedness will influence the effect of the ALAC intervention on participants' physical activity, physical functioning, and program engagement. Hypothesis 3B: Neighborhood characteristics, like walkability, crime rate, air quality, access to green space, and neighborhood social vulnerability, will be related to the effectiveness of the ALAC program in terms of enrollment and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Past diagnosis of invasive cancer, or a caregiver (family or friend) of a participating survivor.
2. No longer receiving treatment for cancer (except hormone therapy or long-term maintenance chemotherapy).
3. Over the age of 18.
4. Screen negative for contraindicating health problems on the adapted Physical Activity Readiness Questionnaire (PAR-Q),79 or screened positive but have approval from a health care provider to participate.
5. Lives in the Acres Homes neighborhood of Houston, Texas or has a home zip code of 77088 or 77091.
6. Able to provide informed consent.

Exclusion Criteria:

1. Women who are pregnant (as indicated by self-report).
2. Has participated in the ALAC program within the past year and attended more than 2 group sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Re-AIM Framework | Through study completion; an average of 1 year.
  1. Physical functioning change from baseline to 12 weeks, as measured by the 30-second sit-to-stand test

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, BA,MPH,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org